CLINICAL TRIAL: NCT00169130
Title: Prospective Study of ACVBP Followed by Autologous Stem Cell Transplantation in Case of BCL-2 Overexpression in Non Previously Treated Patients Aged 60 Years or Less With Low-Intermediate Risk Diffuse Large B-Cell Lymphoma
Brief Title: ACVBP Followed by ASCT in Patients With BCL-2 Positive Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Collaborators: Fondation ARC (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNH98-B2
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-07-13 (Estimated); Status verified 2007-07

CONDITIONS: Lymphoma, Large-Cell, Diffuse
Keywords: lymphoma; autologous stem cell transplant; chemotherapy; BCL2
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — Doxorubicin; Cyclophosphamide

INTERVENTIONS:
Drug: doxorubicin
Drug: cyclophosphamide
Procedure: Autologous stem cell transplantation

SUMMARY:
The primary objective of the study is to evaluate the efficacy of ASCT as consolidation in case of bcl-2 overexpression in non previously treated patients aged 60 years or less with low-intermediate risk diffuse large B-cell lymphoma who responded to ACVBP regimen. Our goal is to obtain a 15% increase of event-free survival at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diffuse large B-cell lymphoma according to the WHO classification (anti CD20 labeling)
* Aged 18 to 60 years
* Non previously treated
* With one and only one of the following adverse characteristics: ECOG performance status 2 or more, or Ann Arbor stage III or IV, or elevated LDH level
* Negative HIV, HBV and HCV serologies (except vaccination)
* With a minimum life expectancy of 3 months
* Having previously signed a written informed consent

Exclusion Criteria:

* Any history of treated or non-treated indolent lymphoma.
* T-cell lymphoma.
* Central nervous system or meningeal involvement by lymphoma.
* Any Contra-indication to any drug contained in the chemotherapy regimens.
* Poor renal function (creatinin level>150µmol/l), poor hepatic function (total bilirubin level>30mmol/l, transaminases>2.5 maximum normal level) unless these abnormalities are related to the lymphoma.
* Serious active disease (according to the investigator's decision).
* Poor bone marrow reserve as defined by neutrophils <1.5G/l or platelets<100G/l, unless related to bone marrow infiltration.
* Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.
* Childbearing woman.
* Patients previously treated with an organ transplantation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300
Dates: Start 1999-10

PRIMARY OUTCOMES:
Event free survival.

SECONDARY OUTCOMES:
Complete response rate at the end of treatment.
Disease-free survival for complete responders.
Overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Morel, MD, Principal Investigator — Centre Hospitalier Schaffner, Lens FRANCE
Locations (5):
- Service d'Hematologie, Mont-Godinne, Belgium
- France (4):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen

REFERENCES:
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In French) — http://www.gela.org